CLINICAL TRIAL: NCT03715153
Title: Efficacy and Safety of Bumetanide Oral Liquid Formulation in Children Aged From 2 to Less Than 7 Years Old With Autism Spectrum Disorder. A 6-month Randomised, Double-blind, Placebo Controlled Multicentre Parallel Group Study to Evaluate Efficacy and Safety of Bumetanide 0.5mg Twice a Day Followed by an Open Label Active 6-month Treatment Period With Bumetanide (0.5mg Twice a Day) and a 6 Weeks Discontinuation Period After Treatment Stop.
Brief Title: Efficacy and Safety of Bumetanide Oral Liquid Formulation in Children Aged From 2 to Less Than 7 Years Old With Autism Spectrum Disorder.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The 6-month efficacy analysis did not show any significant difference between bumetanide versus placebo in the treatment of ASD in the overall studied population. No unexpected safety concerns were identified.
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-95008-002; 2017-004420-30 (EudraCT Number)
Record Dates: First submitted 2018-10-12; First posted 2018-10-23 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Bumetanide

STUDY DESIGN:
Intervention Model Description: 6-month, randomized, double-blind, placebo-controlled, parallel groups followed by an open label active 6-month treatment period with bumetanide.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BUMETANIDE (S95008) followed by Open-Label S95008 (Experimental): Participants will receive S95008 for 6 months, 26 weeks, and then they will begin an open-label 6 month treatment period with S95008.
  Interventions: Drug: BUMETANIDE (S95008) for week 0 - 26; Drug: Open-Label BUMETANIDE (S95008) for weeks 26 - 52
- PLACEBO followed by Open-Label S95008 (Placebo Comparator): Participants will receive placebo for 6 months, 26 weeks, and then they will begin an open-label 6 month treatment period with S95008.
  Interventions: Drug: PLACEBO for week 0 - 26; Drug: Open-Label BUMETANIDE (S95008) for weeks 26 - 52

INTERVENTIONS:
Drug: BUMETANIDE (S95008) for week 0 - 26 — Oral solution dosed at 0.5 mg/mL Taken twice daily.
  Arms: BUMETANIDE (S95008) followed by Open-Label S95008
Drug: PLACEBO for week 0 - 26 — Oral solution Taken twice daily.
  Arms: PLACEBO followed by Open-Label S95008
Drug: Open-Label BUMETANIDE (S95008) for weeks 26 - 52 — Oral solution dosed at 0.5 mg/mL Taken twice daily.

SUMMARY:
The purpose of this study was to evaluate the efficacity and the safety of bumetanide/S95008 in the improvement of Autism Spectrum Disorder core symptoms.

DETAILED DESCRIPTION:
The present study (CL3-95008-002) was performed in children from 2 to less than 7 years old presenting with ASD. A 6-month double-blind treatment period was performed in which efficacy and safety of bumetanide 0.5mg BID were assessed versus placebo. This double-blind period was followed by a 6-month open label treatment period of bumetanide 0.5mg twice daily in which long term safety was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 2 to less than 7
* Primary diagnosis of ASD as per Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria
* Criteria met for ASD on Autism Diagnostic Observation Schedule-Generic (ADOS-2) and Autism Diagnosis Interview Revised (ADI-R)
* CGI (Clinical Global Impression) - Severity rating Score ≥ 4
* Childhood Autism Rating Scale second edition (CARS2-ST or HF) total raw score ≥ 34
* Social responsiveness Scale second edition (SRS-2) total score ≥ 66 T-Score
* Absence of diagnosis of Fragile X or Rett Syndrome
* Absence of any clinically significant abnormality likely to interfere with the conduct of the study according to the judgment of the investigator.

Exclusion Criteria:

* Patients not able to follow the study assessments defined by the protocol, with the exception of self-rating questionnaires which will be assessed by parent/legal representative/caregiver for those patients unable to complete them
* Patients having a high suicidal risk according to the investigator judgement
* Chronic renal dysfunction
* Chronic cardiac dysfunction
* Patient with unstable psychotherapy, behavioural, cognitive or cognitive-behavioural therapy
* Severe electrolyte imbalance that is likely to interfere with the study conduct or evaluation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- Richmond Behavioral Associates, Staten Island, New York, United States
- Australia (2):
  - Liverpool Hospital, Liverpool
  - The Royal Children's Hospital Melbourne, Parkville
- Brazil (6):
  - Trial Tech em Pesquisas com Medicamentos Ltda, Curitiba
  - Hospital Universitário Walter Cantídio-Universidade Federal do Ceará, Fortaleza
  - Clínica Neurológica e Neurocirúrgica de Joinville, Joinville
  - Hospital São Vicente de Paulo, Passo Fundo
  - Universidade Federal de São Paulo, Escola Paulista de Medicina, São Paulo
  - Faculdade de Medicina da Universidade de São Paulo - Departamento de psiquiatra, São Paulo
- Czechia (3):
  - University hospital of Ostrava, Department of Psychiatry, Poruba, Ostrava
  - University Hospital Brno, Department of Child Neurology, Brno
  - Institute of Neuropsychiatric Care, Department of Child Psychiatry, Prague
- France (9):
  - GSC CHU-LENVAL Centre ressource autisme, Nice, Alpes-Maritimes
  - Centre d'Investigation Clinique de Lyon, Bron, Auvergne-Rhône-Alpes
  - Hôpital Le Vinatier CRA Rhône-Alpes, Bat 211, Bron, Auvergne-Rhône-Alpes
  - Hôpitaux Universitaires de Strasbourg Service de Psychiatrie de l'Enfant et de l'Adolescent, Strasbourg, Grand Est
  - CHU Rouen, Rouen, Normandy
  - Centre Hospitalier du Rouvray Centre de Ressources pour l'Autisme, Sotteville-lès-Rouen, Normandy
  - Centre Hospitalier Charles Perrens CRA Aquitaine, Bordeaux, Nouvelle-Aquitaine
  - Hôpital des Enfants-Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Robert Debré Service de Psychiatrie de l'enfant et de l'adolescent, Paris, Île-de-France Region
- Hungary (5):
  - Vadaskert Korhaz es Szakambulancia, Budapest
  - Servus Salvus Kft., Budapest
  - Magyar Református Egyház Bethesda Gyermekkórháza, Budapest
  - Bekes Megyei Kozponti Korhaz Gyermek es ifjusagpszichiatriai osztaly, Gyula
  - Szegedi Tudományegyetem Szent-Gyorgy Albert Klinikai Kozpont Gyermekgyógyászati Klinika Gyermek es Ifjusagpszichiátriai o, Szeged
- Italy (6):
  - Neuro Riabilitazione/Psicopatologia dell'età evolutiva Istituto Scientifico Medea - Bosisio Parini, Bosisio Parini, Lombardy
  - U.O. di Neuropsichiatria Infantile Fondazione Istituto Neurologico Nazionale Casimiro Mondino Istituto di Ricovero e Cura a Carattere Scientifico, Pavia, Lombardy
  - Clinica di Neuropsichiatria dell'Infanzia e dell'Adolescenza Ospedale Pediatrico-Microcitemico, Cagliari, Sardinia
  - Programma Interdipartimentale "Autismo 0-90" A.O.U. Policlinico "Gaetano Martino", Messina, Sicily
  - U.O.C. Psichiatria dello Sviluppo IRCCS Fondazione Stella Maris, Calambrone, Tuscany
  - U.O. di Neuropsichiatria Infantile Azienda Ospedaliera Universitaria Senese, Siena, Tuscany
- Poland (5):
  - "Niepubliczny Zakład Opieki Zdrowotnej Gdańskie Centrum Zdrowia Sp. z o.o., Gdansk
  - Centrum Badań Klinicznych PI-House sp. z o.o, Gdansk
  - NAVICULA Centrum Diagnozy i Terapii Autyzmu w Łodzi, Lodz
  - Fundacja SYNAPSIS ul., Warsaw
  - Samodzielny Publiczny Dziecięcy Szpital Kliniczny w Warszawie Oddział Kliniczny Psychiatrii Wieku Rozwojowego, Warsaw
- Centro Hospitalar e Universitario de Coimbra Hospital Pediatrico, Coimbra, Portugal
- Slovakia (2):
  - National Institute of Children Diseases, Department of Child Psychiatry, Bratislava
  - EPAMED, s.r.o., Košice
- Spain (7):
  - Hospita Mutua de Terrassa, Terrassa, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Niño Jesus, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
- United Kingdom (3):
  - Colchester Hospital, Colchester
  - ReCognition Health, London
  - The Winnicott Centre 195-197 Hathersage Road, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Derived] Hawken N, Falissard B, Choquet C, Francois C, Tardu J, Schmid R. Exit interviews from two randomised placebo-controlled phase 3 studies with caregivers of young children with autism spectrum disorder. Front Child Adolesc Psychiatry. 2024 Jun 5;3:1236340. doi: 10.3389/frcha.2024.1236340. eCollection 2024. PMID 39816573
- [Derived] Fuentes J, Parellada M, Georgoula C, Oliveira G, Marret S, Crutel V, Albarran C, Lambert E, Penelaud PF, Ravel D, Ben Ari Y. Bumetanide oral solution for the treatment of children and adolescents with autism spectrum disorder: Results from two randomized phase III studies. Autism Res. 2023 Oct;16(10):2021-2034. doi: 10.1002/aur.3005. Epub 2023 Oct 4. PMID 37794745
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data] — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The following study periods are presented:
  1. Double-blind period of 6 months (Week 0-Week 26): randomized groups are Bumetanide and Placebo.
  2. Open-label active treatment period (Week 26-Week 52): all patients received Bumetanide.
Period: Double-blind Period (From W0 to W26)
Arm/Group | BUMETANIDE (S95008) Followed by Open-Label S95008 | PLACEBO Followed by Open-Label S95008
Started | 107 | 104
Completed | 90 | 95
Not Completed | 17 | 9
Not completed — Protocol Violation | 1 | 1
Not completed — Non medical reason | 8 | 2
Not completed — Adverse Event | 8 | 6
Period: Open-label Period (From W26 to W52)
Arm/Group | BUMETANIDE (S95008) Followed by Open-Label S95008 | PLACEBO Followed by Open-Label S95008
Started | 86 (Not all participants who completed the double-blind phase chose to continue into the open-label period.) | 92 (Not all participants who completed the double-blind phase chose to continue into the open-label period.)
Completed | 46 | 50
Not Completed | 40 | 42
Not completed — Adverse Event | 8 | 3
Not completed — Non medical reason | 31 | 38
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- BUMETANIDE (S95008) Followed by Open-Label S95008: BUMETANIDE/S95008: Oral solution dosed at 0.5 mg/mL. Taken twice daily from weeks 0-26, followed by open-label S95008 for weeks 26-52.
- PLACEBO Followed by Open-Label S95008: PLACEBO: Oral solution. Taken twice daily from weeks 0-26, followed by open-label S95008 for weeks 26-52.
- Total: Total of all reporting groups
Arm/Group | BUMETANIDE (S95008) Followed by Open-Label S95008 | PLACEBO Followed by Open-Label S95008 | Total
Number analyzed (Participants) | 107 | 104 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 107 | 104 | 211
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.4 (1.2) | 4.6 (1.1) | 4.5 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 89 | 87 | 176
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 8 | 8 | 16
  United States | 2 | 1 | 3
  Czechia | 6 | 6 | 12
  United Kingdom | 11 | 11 | 22
  Portugal | 3 | 3 | 6
  Spain | 16 | 17 | 33
  Brazil | 15 | 15 | 30
  Poland | 14 | 13 | 27
  Italy | 15 | 15 | 30
  Slovakia | 3 | 2 | 5
  Australia | 2 | 2 | 4
  France | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Childhood Autism Rating Scale, Second Edition (CARS2) Total Raw Score
Description: The CARS2 total raw score range from 15 to 60. This scale is a behaviour rating scale intended to diagnose autism. A total score of 15 indicates that an individual behaviour is within normal limits, whereas a value of 60 indicates that the individual's behaviour is severly abnormal.
  In term of change from baseline, the greater the mean value decreases, the better it is.
Time Frame: Change from baseline to Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BUMETANIDE (S95008): BUMETANIDE/S95008: Oral solution dosed at 0.5 mg/mL Taken twice daily.
- PLACEBO: PLACEBO: Oral solution Taken twice daily.
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 107 | 104
score on a scale | -3.66 (4.52) | -3.88 (5.06)
Statistical Analysis 1: Comparison: BUMETANIDE (S95008) vs PLACEBO; Test type: Superiority; p = 0.617, t-test, 2 sided; General Linear Model including the fixed, categorical effects of treatment, country, gender, as well as the continuous, fixed covariates of baseline; Estimate of the adjusted difference = 0.35, 95% CI 2-sided [-1.04 to 1.75], Standard Error of Mean 0.71 — Estimate of the adjusted difference was based on 211 patients (Missing data were imputed)

2. Secondary Outcome: Social Responsiveness Scale, Second Edition (SRS-2) Total Raw Score
Description: The SRS-2 total raw score serves as an index of severity of social deficits in the autism spectrum.
  The total raw score ranges from 65 to 260. A value of 65 represents no symptoms disorders, a value of 260 represents a severe autism spectrum disorder.
  In terms of change from baseline, the greater the mean value decreases, the better it is.
Time Frame: Change from baseline to Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 105 | 104
score on a scale | -16.3 (21.9) | -18.7 (24.8)
Statistical Analysis 1: Comparison: BUMETANIDE (S95008) vs PLACEBO; Test type: Superiority; Estimate of the adjusted difference = 0.48, 95% CI 2-sided [-5.91 to 6.88], Standard Error of Mean 3.26 — General Linear Model including the fixed, categorical effects of treatment, country, gender, as well as the continuous, fixed covariates of baseline. Estimate of the adjusted difference was based on 211 patients (Missing data were imputed)

3. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score
Description: Scale which assesses the severity of the illness and the global improvement of the patient under study treatment.
  It ranges from 1 (normal) through to 7 (amongst the most severely ill patients).
Time Frame: At Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 85 | 89
score on a scale | 2.9 (0.8) | 3.1 (0.9)
Statistical Analysis 1: Comparison: BUMETANIDE (S95008) vs PLACEBO; Test type: Superiority; Estimate of the adjusted difference = -0.04, 95% CI 2-sided [-0.24 to 0.16], Standard Error of Mean 0.10 — Rank-based analysis (Wilcoxon scores) including terms for fixed categorical effects of treatment, country and gender. Estimate of the adjusted difference was based on 211 patients (Missing data were imputed)

4. Secondary Outcome: Vineland Adaptative Behaviour Scale II (VABS II)
Description: Scale designated to measure adaptative behaviour The scale for behaviour ranges from 1 to 67. The more the score decreases, the better it is.
Time Frame: Change from baseline to Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 101 | 95
score on a scale | 1.1 (6.1) | 0.7 (5.3)
Statistical Analysis 1: Comparison: BUMETANIDE (S95008) vs PLACEBO; Test type: Superiority; Estimate of the adjusted difference = 0.16, 95% CI 2-sided [-1.42 to 1.75], Standard Error of Mean 0.81 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Patients With Abnormalities in 12-leads Electrocardiogram (ECG) Parameters
Description: Number of patients with clinically significant ECG abnormalities
  The 12-lead electrocardiogram (ECG) is a medical test that is recorded using leads, or nodes, attached to the body. Electrocardiograms (ECGs), capture the electrical activity of the heart and transfer it to graphed paper where abnormalities are reported and interpretated by the cardiologist.
Time Frame: Week 26
Population: As this measure was collected through week 26, only data gathered during the double-blind period for arms Bumetanide and Placebo were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 78 | 77
Participants | 0 | 0

6. Secondary Outcome: Columbia-Suicide Severity Scale Children's Version (C-SSRS-C)
Description: Number of patients with suicidal ideation or suicidal behavior. The scale is 0 to 5 with the highest suicidal behavior being a 5 and the absence of suicidal behavior or very minor behaviors are 0. However, statistical analysis was done by looking at the number of patients with suicidal behavior or suicidal ideation during their lifetime and during the last 6 months of treatment.
Time Frame: Week 26
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 103 | 101
Participants
  During lifetime: suicidal behavior | 0 | 0
  During lifetime: suicidal ideation | 0 | 0
  During the last 6 months in the study: suicidal behavior | NA — Suicidal behavior was not evaluated during the past 6 months. | NA — Suicidal behavior was not evaluated during the past 6 months.
  During the last 6 months in the study: suicidal ideation | 0 | 1

7. Secondary Outcome: Acceptability and Palatability Questionnaires - Only Descriptive Analyses
Description: Acceptability and palatability criterion Based on your child's reactions (indirect rating), do you think that he/she found the administration method to be
Time Frame: Week 26
Population: Missing values are cancelled
Measure: Count of Participants; unit: Participants
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 99 | 102
Participants
  5 (Very satisfactory) | 53 | 58
  4 (Satisfactory) | 30 | 23
  3 (Acceptable) | 10 | 17
  2 (Not very satisfactory) | 5 | 3
  1 (Not satisfactory) | 1 | 1

8. Secondary Outcome: Paediatric Quality of Life Inventory (PedsQL) Questionnaire
Description: It represents the assessment of parent/legal representative perception of patient health related quality of life The values of the questionnaire range from 0 to 100. Higher scores indicate better HRQOL (Health-Related Quality of Life)
Time Frame: Change from baseline to week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BUMETANIDE (S95008) | PLACEBO
Number analyzed (Participants) | 107 | 104
score on a scale | 5.87 (16.37) | 5.47 (21.41)
Statistical Analysis 1: Comparison: BUMETANIDE (S95008) vs PLACEBO; Test type: Superiority; Estimate of the adjusted difference = -0.26, 95% CI 2-sided [-5.12 to 4.59], Standard Error of Mean 2.48

9. Secondary Outcome: Number of Participants Experiencing at Least 1 Treatment Emergent Adverse Event (TEAE)
Time Frame: through week 52
Population: The overall number of participants analyzed reflects the total number of individual patients analyzed. However, since the statistical analysis of TEAE occurrence was separated by period (double-blind, and open-label) many patients were counted once for each period, and thus the sum of participants in each row is greater than the total number of individual participants analyzed. Not all patients who participated in the double-blind period continued into the open-label period.
Measure: Count of Participants; unit: Participants
Groups:
- BUMETANIDE (S95008) Followed by Open-Label S95008: Participants will receive S95008 for 6 months, 26 weeks, and then they will begin an open-label 6 month treatment period with S95008.
  BUMETANIDE (S95008): Oral solution dosed at 0.5 mg/mL Taken twice daily.
- PLACEBO Followed by Open-Label S95008: Participants will receive placebo for 6 months, 26 weeks, and then they will begin an open-label 6 month treatment period with S95008.
  PLACEBO: Oral solution Taken twice daily.
Arm/Group | BUMETANIDE (S95008) Followed by Open-Label S95008 | PLACEBO Followed by Open-Label S95008
Number analyzed (Participants) | 107 | 104
Participants
  Reported during the double-blind period (Week 0 - 26) | 103 | 96
  Reported during the open-label period (Week 26-52): number analyzed (Participants) | 84 | 92
  Reported during the open-label period (Week 26-52) | 84 | 81

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study until the participant's last study visit, ie 1 year.
Description: During the double blind period, the Treatment Emergent Adverse Events (TEAEs) were analyzed between week 0 and week 26.
  During the open-label period for patients initially randomized in placebo group (Placebo/S95008), TEAEs were analyzed between Week 26 and Week 52 (ie when these patients received bumetanide).
  For patients initially randomized in S950098 group and entering in the open-label period (S95008/S95008), treatment emergent adverse events were analyzed from week 0 to week 52.
Groups:
- S95008 - Double-blind Period (Week 0-26): Patients randomised in the bumetamide arm receiving bumetanide during the double-blind period (Week 0-Week 26)
- Placebo - Double-blind Period (Week 0-26): Patients randomised in the placebo arm receiving placebo during the double blind period (week 0 to week 26)
- S95008/S95008 - Open-Label Extension Period (Week 26-52): Patients initially randomized into the bumetamide arm for the double-blind period (Week 0-Week 26) and during the open-label period (Week 26-week 52)
- Placebo/S95008 - Open-Label Extension Period (Week 26-52): Patients initially randomized into the placebo arm for the double-blind period (Week 0-Week 26) and during the open-label period (Week 26-week 52)
Arm/Group | S95008 - Double-blind Period (Week 0-26) | Placebo - Double-blind Period (Week 0-26) | S95008/S95008 - Open-Label Extension Period (Week 26-52) | Placebo/S95008 - Open-Label Extension Period (Week 26-52)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/104 | 0/84 | 0/92
Serious Adverse Events (participants affected / at risk) | 7/107 | 3/104 | 7/84 | 2/92
Other Adverse Events (participants affected / at risk) | 103/107 | 96/104 | 84/84 | 81/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S95008 - Double-blind Period (Week 0-26) (N=107) | Placebo - Double-blind Period (Week 0-26) (N=104) | S95008/S95008 - Open-Label Extension Period (Week 26-52) (N=84) | Placebo/S95008 - Open-Label Extension Period (Week 26-52) (N=92)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multisystem inflammatory syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Atonic seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S95008 - Double-blind Period (Week 0-26) (N=107) | Placebo - Double-blind Period (Week 0-26) (N=104) | S95008/S95008 - Open-Label Extension Period (Week 26-52) (N=84) | Placebo/S95008 - Open-Label Extension Period (Week 26-52) (N=92)
Blood creatinine increased (Investigations) | 6 (6) | 3 (3) | 11 (11) | 5 (5)
Blood uric acid increased (Investigations) | 5 (6) | 0 (0) | 5 (6) | 2 (2)
Weight decreased (Investigations) | 13 (13) | 2 (2) | 12 (13) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (8) | 6 (7) | 6 (7)
Akathisia (Nervous system disorders) | 8 (8) | 4 (5) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 6 (10) | 2 (2) | 2 (2)
Fatigue (General disorders) | 10 (11) | 2 (2) | 7 (8) | 4 (4)
Pyrexia (General disorders) | 10 (11) | 8 (13) | 13 (19) | 12 (13)
Thirst (General disorders) | 62 (76) | 36 (40) | 50 (66) | 30 (36)
Affect lability (Psychiatric disorders) | 6 (6) | 8 (11) | 5 (5) | 6 (7)
Aggression (Psychiatric disorders) | 7 (8) | 9 (9) | 5 (6) | 7 (7)
Anger (Psychiatric disorders) | 7 (8) | 7 (9) | 6 (8) | 4 (4)
Impulsive behavior (Psychiatric disorders) | 3 (3) | 9 (12) | 3 (3) | 5 (6)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (3) | 6 (6) | 6 (6)
Initial insomnia (Psychiatric disorders) | 6 (6) | 6 (6) | 6 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (10) | 6 (6) | 7 (9) | 3 (3)
Irritability (Psychiatric disorders) | 16 (17) | 16 (19) | 16 (19) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 5 (5) | 8 (11) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (13) | 5 (5) | 15 (18) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 11 (16) | 12 (15) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 20 (27) | 11 (15) | 19 (29) | 9 (9)
Vomiting (Gastrointestinal disorders) | 16 (23) | 15 (19) | 16 (28) | 10 (12)
Pollakiuria (Renal and urinary disorders) | 10 (10) | 5 (5) | 9 (10) | 2 (2)
Polyuria (Renal and urinary disorders) | 39 (46) | 23 (25) | 33 (43) | 26 (27)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 5 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 17 (17) | 16 (18) | 15 (19) | 10 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (29) | 2 (2) | 18 (37) | 21 (35)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 6 (6) | 2 (5) | 4 (9)
Increased appetite (Metabolism and nutrition disorders) | 14 (14) | 10 (15) | 15 (16) | 3 (3)
Polydipsia (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 7 (7) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 9 (9) | 5 (5) | 9 (9) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 5 (6) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (17) | 11 (14) | 16 (27) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 4 (5) | 7 (10) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 6 (7) | 7 (10) | 7 (9) | 5 (6)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 4 (4) | 10 (10) | 5 (5)
Creatinine urine dedreased (Investigations) | 4 (4) | 0 (0) | 6 (7) | 2 (2)
Urine calcium increased (Investigations) | 4 (4) | 1 (1) | 6 (6) | 6 (6)
Hypercalciuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 5 (5) | 2 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Enuresis (Psychiatric disorders) | 4 (4) | 2 (4) | 4 (4) | 4 (5)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 2 (2) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 3 (4)
Rhinitis (Infections and infestations) | 2 (2) | 7 (7) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
The sponsor decided to stop the S95008 development and prematurely discontinue the extension period. This decision was not related to unexpected safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03715153/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03715153/SAP_001.pdf